CLINICAL TRIAL: NCT06668584
Title: A Phase II Open-label Study of Olutasidenib Post-transplant Maintenance Therapy for Patients With IDH1-mutated Myeloid Malignancies
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-0522; NCI-2025-00104 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2024-10-30; First posted 2024-10-31 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Myeloid Malignancies
MeSH Terms: interventions — olutasidenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Olutasidenib Maintenance Therapy (Experimental): Starting 30-120 days post-stem cell infusion, patients receive olutasidenib PO BID on days 1-28 of each cycle. Cycles repeat every 28 days for up to 2 years in the absence of disease progression or unacceptable toxicity. Patients also undergo blood sample collection throughout the study. Additionally, patients may undergo bone marrow aspiration and biopsy, ECHO/MUGA scan and chest x-ray at screening.
  Interventions: Drug: Olutasidenib

INTERVENTIONS:
Drug: Olutasidenib — Given by mouth

SUMMARY:
The goal of this clinical research study is to learn about the safety and tolerability of giving olutasidenib to patients with IDH1-mutated myeloid malignancies as maintenance therapy after they receive a stem cell transplant.

DETAILED DESCRIPTION:
Primary Objective:

To determine the safety and tolerability of olutasidenib as maintenance post-alloSCT.

Secondary Objectives:

I. To determine the rate of progression-free survival (PFS) of patients with IDH1 mutated myeloid malignancies who have undergone a stem cell transplant on olutasidenib post-transplant.

II. To determine response rate, overall survival (OS), cumulative incidence of relapse, non-relapse mortality (NRM), graft versus host disease (GVHD) relapse-free survival (GRFS), rate and grading of acute GVHD (aGVHD) grade 2-4 and 3-4 at day 100, incidence and grading chronic GVHD (cGVHD) all grades.

OUTLINE:

Starting 30-120 days post-stem cell infusion, patients receive olutasidenib orally (PO) twice daily (BID) on days 1-28 of each cycle. Cycles repeat every 28 days for up to 2 years in the absence of disease progression or unacceptable toxicity. Patients also undergo blood sample collection throughout the study. Additionally, patients may undergo bone marrow aspiration and biopsy, echocardiography (ECHO)/multigated acquisition (MUGA) scan and chest x-ray at screening.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of AML, MDS, MPN, or CMML according to World Health Organization (WHO) classification that underwent first or second alloSCT regardless of stem cell source, donor type/match, conditioning regimen, or GVHD prophylaxis and is at least 30 days post stem cell transplant until day 120.
2. Evdence of an IDH1 mutation presence by next generation sequencing panel at original diagnosis.
3. Evidence of engraftment by Absolute neutrophil count (ANC) >/= 1.0x 109/L without daily use of myeloid growth factor (G-CSF) for at least 7 days; and Platelet >/= 30 x 109/L with out platelet transfusion within 1 week.
4. Patient in morphologic remission with Day +30 bone marrow <5% blast. Will include MRD positive or negative.
5. Age 18 to 75 years old.
6. ECOG performance status of 0, 1, 2. Or KPS above 70.
7. Creatinine clearance greater or equal to 40cc/min as defined by the Cockcroft-Gault Equation.

   Males (mL/min): (140-age) *IBW (kg) / 72*(serum creatinine(mg/dl)) Females (mL/min): 0.85*(140-age) *IBW (kg) / 72*(serum creatinine(mg/dl)).
8. Serum bilirubin </= 1.5 x upper limit of normal (ULN) except in subjects with Gilbert's Syndrome in whom total bilirubin must be </= 3.0 mg/dl. Aspartate transaminase (AST) or alanine transaminase (ALT) </= 2.5 x ULN. Alkaline phoshatase </=2.5 x ULN.
9. No active bleeding.
10. No clinical evidence of life-threatening infection.
11. Capable of understanding the investigational nature, potential risks, and benefits of the study, and able to provide valid informed consent.
12. Negative serum or urine pregancy test for wome with reproductive potential at screening.
13. Female participants of non-childbearing potential must meet at least one of the following criteria:

    1. Postmenopausal (no menses in greater than or equal to 12 consecutive months).
    2. History of hysterectomy or bilateral salpingo-oophorectomey.
    3. Ovarian failure (follicle-stimulating hormone and Estradiolin menopausal range, who have received Whole Pelvic Radiation Therapy).
    4. History of bilateral tubal ligation or another surgical sterilization procedure
14. Subjects who are of childbearing potential, sexually active, and at risk of pregnancy must agree to use a highly effective method of contraception for the duration of the active treatment and at least 3 months post-completion of the study therapy. See Appendix B.

Approved methods of birth control are as follows: Hormonal contraception (i.e., birth control pills, injection, implant, transdermal patch, vaginal ring), Intrauterine device (IUD), Tubal Ligation or hysterectomy, Subject/Partner post vasectomy, Implantable or injectable contraceptives, and condoms plus spermicide. Not engaging in sexual activity for the total duration of the trial and the drug washout period is an acceptable practice however periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. See Appendix B.

Men treated or enrolled in this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of Olutasidenib administration.

Exclusion Criteria:

1. Use of any of the following after transplantation and prior to starting study therapy. Anti-leukemic agents given as post-transplant maintenance therapy (e.g., subcutaneous, or oral 5-azacitidine or FL T3 inhibitors for maintenance)
2. Overall grade II-IV aGVHD. However, upon complete resolution of aGVHD-related symptoms with grade 1 or 0 overall clinical grade would be appropriate to enroll at that time. Patients may be eligible for enrollment if they are on prednisone 0.5 mg/kg daily dose or lower, tacrolimus, sirolimus, and/or ruxolitinib.
3. cGVHD, moderate or servere by NIH criteria.
4. Active uncontrolled systemic fungal, bacterial, or viral infection. However, patients receiving anti-micobial agents including antibiotics, antiviral and antifungal therapies are allowed if the infection is controlled, and the patient is hemodynamically stable.
5. Known active viral infection with Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV), or Hepatitis C Virus (HCV).

   * Patients with known active hepatitis B virus (HBV) infection will be excluded because of potential effects on immune function and/or drug interactions. However, if a patient has HBV history with an undetectable HBV load by polymerase chain reaction (PCR), no liver-related complications, and is on definitive HBV therapy that is not contraindicated in this study, then they would be eligible for study.
   * Patients with known active hepatitis C virus (HCV) infection will be excluded because of potential effects on immune function and/or drug interactions. However, if a patient with a history of HCV infection has received definitive therapy (and is now HCV viral load negative), or if a patient has a reactive HCV antibody test but has an undetectable viral load by PCR, then they would be eligible.
   * Patients with known active HIV infection will be excluded out of concern for the drug-drug interaction with venetoclax and highly active antiretroviral therapy (HART)
6. QT prolongation of corrected QTcF interval (QTc) > 480 milliseconds
7. Any other condition that would, in the Investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns with clinical study procedures.
8. Patients with cognitive impairments or psychiatric disorders that can interfere with safety or with obtaining informed consent of compliance with study procedures.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2024-12-31 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Ramdial, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org